CLINICAL TRIAL: NCT03387111
Title: QUILT-3.090: NANT Squamous Cell Carcinoma (SCC) Vaccine: Molecularly Informed Integrated Immunotherapy Combining (haNK) Cell Therapy With Adenoviral and Yeast-based Vaccines to Induce T-cell Responses in Subjects With SCC Who Have Progressed on or After Platinum-based Chemotherapy and Anti-programmed Cell Death Protein 1 (PD-1)/Programmed Death-ligand 1 (PD-L1) Therapy
Brief Title: QUILT-3.090: NANT Squamous Cell Carcinoma (SCC) Vaccine: Subjects With SCC Who Have Progressed
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.090
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2020-08

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — yeast-CEA vaccine; avelumab; Bevacizumab; Capecitabine; Cetuximab; Cisplatin; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; necitumumab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT Squamous Cell Carcinoma (SCC) Vaccine (Experimental): Combination of agents were administered in this study: Aldoxorubicin HCl, ETBX-011, ETBX-021, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, haNK, N-803, avelumab, bevacizumab, capecitabine, cetuximab, cisplatin, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, necitumumab, SBRT.
  Interventions: Drug: Aldoxorubicin HCl; Biological: ETBX-011; Biological: ETBX-021; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6207; Biological: GI-6301; Biological: haNK for infusion; Drug: Avelumab; Drug: bevacizumab; Drug: Capecitabine; Drug: Cetuximab; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Fluorouracil; Drug: Leucovorin; Drug: nab-Paclitaxel; Drug: Necitumumab; Procedure: SBRT; Biological: N-803

INTERVENTIONS:
Drug: Aldoxorubicin HCl — Aldoxorubicin hydrochloride
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
Biological: ETBX-021 — Ad5 [E1-, E2b-]-HER2
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury vaccine
Biological: ETBX-061 — Ad5 [E1-, E2b-]-MUC1
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
Biological: GI-6207 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant CEA proteins
Biological: GI-6301 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Brachyury yeast proteins
Biological: haNK for infusion — NK-92 [CD16.158V, ER IL-2]
Drug: Avelumab — Recombinant human anti-PD-L1 IgG1 monoclonal antibody
Drug: bevacizumab — Recombinant human anti-VEGF IgG1 monoclonal
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Drug: Cetuximab — Cetuximab is an epidermal growth factor receptor (EGFR) antagonist.
Drug: Cisplatin — cis-diamminedichloroplatinum(II)
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
Drug: nab-Paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
Drug: Necitumumab — Necitumumab is a recombinant human lgG1 monoclonal antibody.
Procedure: SBRT — Stereotactic Body Radiation Therapy
Biological: N-803 — Recombinant human superagonist interleukin-15 (IL-15) complex [also known as IL-15N72D:IL-15RuSu/IgGI Fe complex1)
  Other Names: Formerly known as ALT-803

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with SCC who have progressed on or after previous platinum-based chemotherapy and anti-PD-1/PD-L1 therapy. Phase 2 will be based on Simon's two-stage optimal design.

DETAILED DESCRIPTION:
Treatment will be administered in 2 phases, an induction and a maintenance phase, as described below. Subjects will continue induction treatment for up to 1 year. Treatment in the study will be discontinued if the subject experiences progressive disease (PD) or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects who experience ongoing stable disease (SD) or an ongoing partial response (PR) at 1 year may enter the maintenance phase at the Investigator's and Sponsor's discretion. Subjects may remain in the maintenance phase of the study for up to 1 year. The duration of the maintenance phase can exceed 1 year if the subject continues to benefit, per the Investigator's and Sponsor's discretion. Treatment will continue in the maintenance phase until the subject experiences PD or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. The time on study treatment, including both the induction and maintenance phases, is up to 2 years. The duration of the study may exceed 2 years if the subject remains in the maintenance phase for more than 1 year, as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed HNSCC or squamous NSCLC with progression on or after platinum-based chemotherapy and anti-PD-1/PD-L1 therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, or autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count < 1,000 cells//mm^3.
   2. Uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
   3. Platelet count < 75,000 cells/mm^3.
   4. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   8. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Serious myocardial dysfunction defined by ECHO as absolute left ventricular ejection fraction (LVEF) 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 30 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
  Eligible participants could have gone through both induction and maintenance treatment on study.
Period: Overall Study
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Started | 4
Completed | 0
Not Completed | 4
Not completed — Progressive Disease | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- NANT Squamous Cell Carcinoma (SCC) Vaccine: Combination of agents will be administered in this study: Aldoxorubicin HCl, ETBX-011, ETBX-021, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, haNK, N-803, avelumab, bevacizumab, capecitabine, cetuximab, cisplatin, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, necitumumab, SBRT.
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Subjects with SCC who have progressed [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Time Frame: 30 days after last dose, up to 15.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Objective Response Rate by RECIST Version 1.1
Description: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase by computed tomography (CT) or magnetic resonance imaging (MRI) of target and non-target lesions in accordance with RECIST Version 1.1.
  An objective response is defined as a confirmed complete or partial overall response with confirmation occurring at least 4 weeks after the initial response is observed.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression, up to 11 months.
Population: No participants had either confirmed partial response or complete response on study. Therefore, objective response rate is 0.
Measure: Count of Participants; unit: Participants
Groups:
- NANT Squamous Cell Carcinoma (SCC) Vaccine: Combination of agents were administered in this study:
  Aldoxorubicin hydrochloride
  ETBX-011: Ad5 [E1-, E2b-]-CEA
  ETBX-021: Ad5 [E1-, E2b-]-HER2
  ETBX-051: Ad5 [E1-, E2b-]-Brachyury vaccine
  ETBX-061: Ad5 [E1-, E2b-]-MUC1
  GI-4000: Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
  GI-6207: Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant CEA proteins
  GI-6301: Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Brachyury yeast proteins
  haNK for infusion: NK-92 [CD16.158V, ER IL-2]
  Avelumab
  bevacizumab
  Capecitabine
  Cetuximab
  Cisplatin
  Cyclophosphamide
  Fluorouracil: 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Leucovorin
  nab-Paclitaxel
  Necitumumab
  SBRT: Stereotactic Body Radiation Therapy
  N-803: Recombinant human superagonist interleukin-15 (IL-15) complex [also known as IL-15N72D:IL-15RuSu/IgGI Fe complex1)
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: Objective Response Rate by irRC
Description: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase by computed tomography (CT) or magnetic resonance imaging (MRI) of target and non-target lesions in accordance with immune-related response criteria (irRC).
  An objective response is defined as a confirmed complete or partial overall response with confirmation occurring at least 4 weeks after the initial response is observed.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until confirmed disease progression, up to 11 months.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: Progression Free Survival by RECIST Version 1.1.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions PFS was evaluated using Kaplan-Meier methods. PFS was defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first. Subjects completing study follow-up or initiating a new anticancer therapy prior to documented PD was censored in the PFS analysis at the last known date the subject was progression free prior to completing follow-up or initiating the new therapy.
Time Frame: Tumors were assessed at screening, and tumor response was assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression or death (any cause) whichever occurred first, up to 11 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Months | 5.3 [0.8 to NA] — NA = 95% Confidence Interval upper limit was not calculable due to an insufficient number of participants with events

5. Secondary Outcome: Progression Free Survival by irRC
Description: PFS was evaluated using Kaplan-Meier methods. PFS was defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first. Subjects completing study follow-up or initiating a new anticancer therapy prior to documented PD was censored in the PFS analysis at the last known date the subject was progression free prior to completing follow-up or initiating the new therapy.
Time Frame: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Months | 5.7 [4.9 to NA] — NA = 95% Confidence Interval upper limit was not calculable due to an insufficient number of participants with events

6. Secondary Outcome: Overall Survival
Description: OS was evaluated using Kaplan-Meier methods. OS was defined as the time from the date of first treatment to the date of death (any cause). Participants who were alive at the end of follow-up were censored in the OS analysis at the last known date alive.
Time Frame: Participants were assessed from screening to death.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Months | 15.1 [6.4 to NA] — NA = 95% Confidence Interval upper limit was not calculable due to an insufficient number of participants with events

7. Secondary Outcome: Duration of Response (DOR) by RECIST Version 1.1 and irRC
Description: DOR was defined as the time from the date of first response (PR or CR) to the date of disease progression or death (any cause) whichever occurred first. Responding subjects completed study follow-up or initiated a new anticancer therapy prior to documented PD was censored in the DOR analysis at the last known date the subject was progression free prior completing follow-up or initiating the new therapy.
Time Frame: as for outcome 4
Population: There were no participants with confirmed CR or PR. Therefore, no participants were included in the DOR analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Participants | 0

8. Secondary Outcome: Disease Control Rate (Confirmed Complete Response, Partial Response, or Stable Disease Lasting for at Least 2 Months) by RECIST Version 1.1
Description: Disease control is defined as subjects with a confirmed CR, PR, or SD lasting for at least 2 months
Time Frame: Up to 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Participants
  Confirmed Complete Response | 0
  Confirmed Partial Response | 0
  Unconfirmed Complete Response | 0
  Unconfirmed Partial Response | 1
  Stable Disease | 1
  Progressive Disease | 1
  Imaging Not Available to Evaluate | 1

9. Secondary Outcome: Quality of Life (QoL) by Patient Reported Outcomes
Description: QoL was conducted via PROs using the Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) or Functional Assessment of Cancer Therapy - Lung (FACT-L) questionnaire. The FACT-H&N and FACT-L compilation of general questions divided into five QoL subscales: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Additional Concerns.
  It uses 5-point Likert-type response categories ranging from 0 = 'not at all' to 4 = 'very much'. Each subscale consists of 6-12 questions to answer.
Time Frame: Up to 15.5 months
Population: There were 2 QOLs planned on study, FACT-L/FACT-H&N. No participants took the FACT-L. There is no data to summarize. The FACT H&N was performed during the study for 1 participant. The only other participant who took the FACT-H&N performed this QOL at screening only. There is no QOL data to summarize.
  According to the approved SAP, FACT-H&N/FACT-L scores at baseline and post-baseline time points were to be presented in a data listing. The results of the PRO were not planned to be summarized.
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 0

10. Secondary Outcome: Disease Control Rate (Confirmed Complete Response, Partial Response, or Stable Disease Lasting for at Least 2 Months) by irRC
Description: Disease control is defined as subjects with a confirmed CR, PR, or SD lasting for at least 2 months
Time Frame: Up to 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
Number analyzed (Participants) | 4
Participants
  Confirmed irCR | 0
  Confirmed irPR | 0
  Unconfirmed irCR | 0
  Unconfirmed irPR | 1
  irSD | 2
  Unconfirmed irPD | 0
  Confirmed irPD | 0
  Imaging not available to evaluate | 1

ADVERSE EVENTS:
Time Frame: Non-serious AEs were followed for 30 days after the subject's last dose of study treatment, up to 15.5 months. Non-serious grade 3 or 4 AEs were followed until resolution or stabilization, up to 15.5 months. All SAEs that had not resolved upon discontinuation of the subject's participation in the study were followed until recovered, recovered with sequelae, not recovered (death due to other cause), death (due to the SAE), lost to follow-up.
Arm/Group | NANT Squamous Cell Carcinoma (SCC) Vaccine
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Squamous Cell Carcinoma (SCC) Vaccine (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Squamous Cell Carcinoma (SCC) Vaccine (N=4)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 4
Chills (General disorders) | 3
Injection site reaction (General disorders) | 3
Face oedema (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Asthenia (General disorders) | 1
Catheter site pain (General disorders) | 1
Extravasation (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Weight decreased (Investigations) | 3
Blood pressure increased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Conjunctivitis (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Catheter site cellulitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Dry eye (Eye disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Anxiety (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT03387111/Prot_SAP_000.pdf